CLINICAL TRIAL: NCT00349661
Title: Influence Of Omeprazole On The Anti-Platelet Action Of Clopidogrel Associated To Aspirin: Double-Blind Randomized Trial Against Placebo
Brief Title: Influence Of Omeprazole On The Anti-Platelet Action Of Clopidogrel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCLA
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Heart Disease
Keywords: clopidogrel; omeprazole
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Drug: impact on VASP test

SUMMARY:
Objectives: A prospective investigation of the effect of omeprazole, a proton pump inhibitor, on the anti-platelet action of clopidogrel.

The main decision criterion will concern change in VASP protein phosphorylation under treatment. Phosphorylation will be measured before and after administration of omeprazole versus placebo in patients undergoing clopidogrel treatment.

Type of study: Single center, double blind, randomized parallel group study versus placebo, comparing two treatment groups:

* clopidogrel + omeprazole + standard regime (beta-blockers, atorvastatin, IEC, aspirin)
* clopidogrel + placebo+ standard regime (beta-blockers, atorvastatin, IEC, aspirin)

Study population: 120 patients from the Cardiology Department of Brest University hospital, Brest (France), receiving a standard treatment comprising a loading dose of clopidogrel followed by a daily dose of 75 mg associated to 75 mg aspirin, will be randomized between 20 mg/day omeprazole and 20 mg/day placebo treatment groups. The efficacy of clopidogrel will be assessed by inter-group comparison on the VASP test.

Study period: 7 days' treatment per patient. Total study period estimated at 6 months.

Expected findings: The results should confirm the suspected negative effect of omeprazole on clopidogrel's impact on arterial thrombosis risk, secondarily allowing new recommendations to be drawn up for this association.

DETAILED DESCRIPTION:
Preventing recurrence of thrombosis following angioplasty relies on dual-therapy associating the anti-platelet agents aspirin and clopidogrel. This regime is kept up for between 1 and 6 months, depending on the type of stent deployed in the angioplasty. The biological effectiveness of the clopidogrel treatment can be assessed by the VASP test, a new platelet test, results on which have been shown to correlate with risk of thrombosis. A study we ran recently strongly suggested that omeprazole was associated with a poor response to clopidogrel. Omeprazole is an anti-ulcer agent frequently prescribed to prevent unwanted side-effects of aspirin, making it frequently associated to clopidogrel in the aftermath of angioplasty.

Study population: 120 patients from the Cardiology Department of Brest University hospital, Brest (France), receiving a standard treatment comprising a loading dose of clopidogrel followed by a daily dose of 75 mg associated to 75 mg aspirin, will be randomized between 20 mg/day omeprazole and 20 mg/day placebo treatment groups. The efficacy of clopidogrel will be assessed by inter-group comparison on the VASP test.

Study period: 7 days' treatment per patient. Total study period estimated at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patient with indication of aspirin and clopidogrel treatment

Exclusion Criteria:

* patient<18 years
* liver disease
* drug eluting stent
* gastrointestinal ulcus
* bleeding
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
inter group comparison of VASP test

CONTACTS AND LOCATIONS:
Overall Officials: martine gilard, md, Principal Investigator — PI
Locations (1):
- Department of Cardiology, Brest, France

REFERENCES:
- [Derived] Gilard M, Arnaud B, Cornily JC, Le Gal G, Lacut K, Le Calvez G, Mansourati J, Mottier D, Abgrall JF, Boschat J. Influence of omeprazole on the antiplatelet action of clopidogrel associated with aspirin: the randomized, double-blind OCLA (Omeprazole CLopidogrel Aspirin) study. J Am Coll Cardiol. 2008 Jan 22;51(3):256-60. doi: 10.1016/j.jacc.2007.06.064. PMID 18206732